CLINICAL TRIAL: NCT04300777
Title: Clinical Evaluation of the SeaSpine Non-Cervical Pedicle Screw Systems
Brief Title: The Fixation Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: SeaSpine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SS-PMCF-1905
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Degenerative Conditions, Neurologic
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Treated with Non-Cervical Pedicle Screw Systems: 50 patients who have been implanted with SeaSpine Non-Cervical Pedicle Screw Systems
  Interventions: Device: SeaSpine Non-Cervical Pedicle Screw Systems

INTERVENTIONS:
Device: SeaSpine Non-Cervical Pedicle Screw Systems — Any patient treated with a SeaSpine Non-Cervical Pedicle Screw System

SUMMARY:
To perform a clinical evaluation of safety and performance for the SeaSpine Non- Cervical Pedicle Screw Systems

DETAILED DESCRIPTION:
A multi-center, post-market, clinical evaluation for subjects implanted with the SeaSpine Non-Cervical Pedicle Screw Systems

ELIGIBILITY:
Inclusion Criteria:

* Have undergone surgery
* Have undergone at least 12-months of postoperative follow-up

Exclusion Criteria:

* Any condition that the Investigator determines is unacceptable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been implanted with a SeaSpine Non-Cervical Pedicle Screw System
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for the study is device performance. | 12 months post-operative
  Device performance is defined as lack of component failure involving screw and/or rod fracture and/or screw loosening or disassociation.

SECONDARY OUTCOMES:
Evaluation of unanticipated adverse device effects (UADE) | 12-months
  Intra or Post-Procedure UADEs

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vizesi, Ph.D., Study Director — SeaSpine, Inc.
Locations (2):
- United States (2):
  - Henry Ford, Jackson, Michigan
  - OrthoNeuro, New Albany, Ohio